CLINICAL TRIAL: NCT05040386
Title: Nurse Coach-Led Early Palliative Care for Older Adults With Chronic Obstructive Pulmonary Disease and Their Care Partners: The Project EPIC Pilot Randomized Controlled Trial
Brief Title: Nurse Coach-Led Early Palliative Care for Older Adults With COPD and Their Care Partners: The Project EPIC Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anand Iyer, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-300007901; K76AG064327 (NIH)
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: COPD
Keywords: palliative care; supportive care; caregiver; geriatrics; telehealth; chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patient participants randomized to this arm will receive the standard of care for COPD. Caregiver participants, if available, will be randomized to the same study arm as the patient participant.
  Interventions: Other: Usual Care
- Intervention (EPIC) (Experimental): Participants randomized to this arm will receive the experimental treatment for COPD (i.e. EPIC). Caregiver participants, if available, will be randomized to the same study arm as the patient participant.
  Interventions: Behavioral: EPIC (Empower People to Independence in COPD)

INTERVENTIONS:
Behavioral: EPIC (Empower People to Independence in COPD) — EPIC (Empower People to Independence in COPD) is a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. EPIC includes weekly (6 for patients and 4 for caregivers) telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention.
  Arms: Intervention (EPIC)
Other: Usual Care — Participants randomized to this arm receive standard of care for COPD. This includes routine clinic visits with their clinician, medications, inhalers, vaccinations, tobacco cessation counseling, illness education, cardiopulmonary rehabilitation, specialist referrals, and other COPD therapies deemed appropriate by their clinician. Caregiver participants are randomized to the same study arm as the patient participant.
  Arms: Usual Care

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death in older Americans. COPD increases in frequency with age, and older adults with COPD often have significant unmet geriatrics-palliative care needs that results in reduced quality of life, high healthcare utilization, and care at the end of life that does not align with the values and wishes of patients and their care partners. Older adults with COPD could benefit from proactive geriatrics-palliative care before the end of life. However, no geriatrics-palliative care interventions have been systematically developed and tested in community-dwelling older adults with COPD and their care partners. As the number of older adults with COPD increases to levels unmatched by current palliative care workforce trends, innovative strategies are desperately needed to improve the delivery of geriatrics-palliative care in COPD before the end of life.

Project EPIC (Empowering People to Independence in COPD) is a multiphase study to refine and pilot test the EPIC telephonic nurse coaching intervention in older adults with COPD and their care partners. EPIC is informed by the ENABLE (Educate, Nurture, Advise Before Life Ends) early palliative care intervention that improved quality of life and mood for patients with advanced cancer and has been iteratively refined over decades and rigorous randomized controlled trial testing. In the intervention, palliative care-trained nurse coaches deliver the Charting Your Course Curriculum over the phone to patients (six sessions) and their care partners (four sessions), with activities and monthly telephone follow-up following a manualized curriculum. We conducted a formative evaluation in a diverse and multidisciplinary group of stakeholders to refine ENABLE for patients with COPD and pilot tested the potential feasibility of the refined intervention, EPIC, in patients and their care partners.

The current study summatively evaluates EPIC through a hybrid effectiveness-implementation pilot randomized controlled trial in dyads of community-dwelling older adults with moderate to very severe COPD and their care partners randomized to usual care (control) versus EPIC (intervention). The primary outcomes are intervention feasibility and acceptability. Secondary outcomes include Life-Space mobility, quality of life, cognitive impairment, functional status, palliative care uptake, and care partner burden.

ELIGIBILITY:
Patients

Inclusion criteria (must meet ALL of the following):

1. ≥60 years;
2. COPD on routinely collected spirometry (FEV1/FVC <0.70 + FEV1<80%);
3. Able to speak English;
4. At least one of the following:

4a) Severe breathlessness as defined by a documented modified Medical Research Council (mMRC) Dyspnea Scale Score >2 in the medical record or any of the following levels of severe breathlessness by medical review: breathless after walking about 100 yards, breathless after a walking few minutes on level ground, or too breathless to leave the house or when dressing); OR, 4b) ≥1 hospitalization in the year prior but >30 days from enrollment; OR, 4c) On supplemental oxygen (exertional or continuous).

Exclusion criteria (can be excluded for ANY of the following):

1. No access to a dedicated telephone service;
2. Recent hospitalization for any reason or exacerbation of COPD in the past 30 days or ongoing exacerbation symptoms requiring treatment with antibiotics and steroids;
3. Treated within the past 60 days for an advanced cancer defined as metastatic and/or recurrent/progressive stage III/IV cancer, including brain, lung, breast, gynecologic, head and neck, gastrointestinal, genitourinary cancer, and hematologic malignancies by self report or chart review;
4. Active schizophrenia, major depressive disorder, bipolar disorder, suicidal ideations, or substance abuse by self-report or chart review (Active means currently being treated for schizophrenia, bipolar disorder, or suicidal ideations or having active and untreated major depressive disorder, i.e. not under the care of a clinician or not on medications such as antidepressants or mood stabilizers, or having active and untreated substance abuse, i.e. not on medication or enrolled in a substance abuse program);
5. Non-correctable hearing impairment (i.e. hearing impairment despite hearing aids);
6. Severe cognitive impairment (score ≤3 points on 6-item Callahan Screener): a) Correctly identify current year (1 point); b) Correctly identify current month (1 point); c) Correctly identify current day (1 point); d) Correctly recall "apple" after 5 minutes (1 point); e) Correctly recall "table" after 5 minutes (1 point); f) Correctly recall "penny" after 5 minutes (1 point).

Care partners

Inclusion criteria (must meet ALL of the following):

1. ≥18 years;
2. Self-reporting as "an unpaid spouse or care partner, relative, or friend who knows [the patient] well and is involved in their medical care";
3. Able to speak English.

Exclusion criteria (can be excluded for ANY of the following):

1. No access to a dedicated telephone service;
2. Active schizophrenia, major depressive disorder, bipolar disorder, suicidal ideation, or substance abuse by self-report (Active schizophrenia, major depressive disorder, bipolar disorder, suicidal ideation, or substance abuse by self-report or chart review (Active means currently being treated for schizophrenia, bipolar disorder, or suicidal ideations or having active and untreated major depressive disorder, i.e. not under the care of a clinician or not on medications such as antidepressants or mood stabilizers, or having active and untreated substance abuse, i.e. not on medication or enrolled in a substance abuse program);
3. Non-correctable hearing impairment (i.e. hearing impairment despite hearing aids);
4. Severe cognitive impairment (score ≤3 points on a 6-item Callahan screener): a) Correctly identify current year (1 point); b) Correctly identify current month (1 point); c) Correctly identify current day (1 point); d) Correctly recall "apple" after 5 minutes (1 point); e) Correctly recall "table" after 5 minutes (1 point); f) Correctly recall "penny" after 5 minutes (1 point)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byun JY, Wells R, Bechthold AC, Coffee-Dunning J, Armstrong M, Taylor R, O'Hare L, Dransfield MT, Brown CJ, Vance DE, Odom JN, Bakitas M, Iyer AS. Project EPIC (Empowering People to Independence in COPD): Study protocol for a hybrid effectiveness-implementation pilot randomized controlled trial of telephonic, geriatrics-palliative care nurse-coaching in older adults with COPD and their family caregivers. Contemp Clin Trials. 2024 May;140:107487. doi: 10.1016/j.cct.2024.107487. Epub 2024 Mar 6. PMID 38458558

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (EPIC + Usual Care): Patient Participants: Patient participants randomized to the intervention arm receive the patient-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, alongside usual COPD care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. The patient-focused EPIC intervention includes six once weekly telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention with four caregiver-tailored nurse-coach sessions, instead of six sessions.
- Control (Usual Care): Patient Participants: Participants randomized to this arm receive standard of care for COPD. This includes routine clinic visits with their clinician, medications, inhalers, vaccinations, tobacco cessation counseling, illness education, cardiopulmonary rehabilitation, specialist referrals, and other COPD therapies deemed appropriate by their clinician.
- Intervention (EPIC + Usual Care): Caregiver Participants: Caregiver participants randomized to the intervention arm alongside the patient participant receive the caregiver-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults and their caregivers. The caregiver-focused EPIC intervention includes four once weekly telephone-based, nurse coach-led sessions tailored to caregivers of patients with COPD aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions and complete an Advance Directive.
- Control (Usual Care): Caregiver Participants: Participants randomized to this arm will receive usual care.
Period: Overall Study
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Started | 15 | 15 | 10 | 10
Completed | 14 | 15 | 8 | 10
Not Completed | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention (EPIC + Usual Care): Patient Participants: Patient participants randomized to the intervention arm receive the patient-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, alongside usual care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. The patient-focused EPIC intervention includes six once weekly telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention with four caregiver-tailored nurse-coach sessions, instead of six sessions.
- Total: Total of all reporting groups
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants | Total
Number analyzed (Participants) | 15 | 15 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.6) | 71.1 (8.1) | 64.3 (15.8) | 62.6 (6.1) | 67.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 8 | 9 | 32
  Male | 10 | 5 | 2 | 1 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 4 | 1 | 14
  White | 9 | 12 | 6 | 9 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 10 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility
Description: In participants randomized to the intervention arm, we will measure the mean (SD) number of core EPIC patient and caregiver telephonic nurse coaching sessions out of a possible 10 and 8 sessions completed, respectively.
Time Frame: 6 months
Population: This sample represents the total patient and caregiver participants who started the EPIC intervention and completed at least the introductory session.
Measure: Mean (Standard Deviation); unit: Sessions
Groups:
- Intervention (EPIC + Usual Care): Participants randomized to the intervention arm receive the EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention for patients with COPD and their caregivers informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, alongside usual COPD care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. The patient-focused EPIC intervention includes six once weekly telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention with four caregiver-tailored nurse-coach sessions, instead of six sessions.
Arm/Group | Intervention (EPIC + Usual Care)
Number analyzed (Participants) | 24
Sessions
  Mean (SD) Patient Core EPIC Sessions: number analyzed (Participants) | 15
  Mean (SD) Patient Core EPIC Sessions | 9.2 (2.4)
  Mean (SD) Caregiver Core EPIC Sessions: number analyzed (Participants) | 9
  Mean (SD) Caregiver Core EPIC Sessions | 6.4 (2.7)

2. Primary Outcome: Survey Feasibility
Description: Survey completion rates will be measured and presented as the count of patient and caregiver participants who completed 100% of all available survey sets across the study.
Time Frame: 6 months
Population: Patient and caregiver participants by study arms are analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention (EPIC): Patient Participants: Patient participants randomized to the intervention arm receive the patient-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. The patient-focused EPIC intervention includes six once weekly telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention with four caregiver-tailored nurse-coach sessions, instead of six sessions.
- Intervention (EPIC): Caregiver Participants: Caregiver participants randomized to the intervention arm alongside the patient participant receive the caregiver-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults and their caregivers. The caregiver-focused EPIC intervention includes four once weekly telephone-based, nurse coach-led sessions tailored to caregivers of patients with COPD aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions and complete an Advance Directive.
Arm/Group | Intervention (EPIC): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 15 | 15 | 10 | 10
Participants | 12 | 12 | 6 | 8

3. Primary Outcome: Intervention Acceptability Score
Description: Mean (SD) score on a scale of 1 being very poor and 10 being excellent for the EPIC intervention as rated by patient and caregiver participants randomized to the intervention group.
Time Frame: 6 months
Population: This represents patient and caregiver participants separately who completed this survey.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Intervention (EPIC + Usual Care): Patient Participants: Patient participants randomized to the intervention arm receive the patient-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. The patient-focused EPIC intervention includes six once weekly telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention with four caregiver-tailored nurse-coach sessions, instead of six sessions.
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants
Number analyzed (Participants) | 13 | 8
Score on a Scale | 9.8 (0.4) | 9.9 (0.4)

4. Primary Outcome: Count of Acceptability Qualitative Interviews
Description: Count of patient and caregiver participants completing the follow-up semi-structured, in-depth interviews.
Time Frame: 6 months
Population: Count of patient and caregiver participants completing the follow-up semi-structured, in-depth interviews.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (EPIC): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 15 | 15 | 10 | 10
Participants | 12 | 12 | 6 | 7

5. Secondary Outcome: UAB Life Space Assessment
Description: The UAB Life Space Assessment is a 15-item measure of Life-Space mobility, or the frequency, distance, and independence of movement in the 4 weeks prior to administration. Scores range from 0 (lowest) to 120 (best), and lower scores are associated with more restricted Life-Space mobility. A threshold score of >=60 is used to identify restricted Life-Space mobility, which is a marker of social isolation, frailty, and predictor of healthcare utilization in older adults. MCID=5 points with an alpha=0.80.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 14 | 14 | 8 | 10
Units on a Scale | 46.6 (20.3) | 52.1 (29.1) | 100.5 (21.9) | 90.3 (17.6)

6. Secondary Outcome: Chronic Respiratory Questionnaire (CRQ)
Description: The Chronic Respiratory Questionnaire (CRQ) is a 20-item measure of quality of life along 4 domains: CRQ dyspnea, CRQ fatigue, CRQ mastery, and CRQ emotional function. Each domain score ranges from 1 (most severe impairment) to 7 (no impairment). Higher scores are better on each domain, with MCID of 0.5 points and an alpha=0.70. The CRQ Dyspnea Domain has a range of 1 to 7, with higher scores associated with a better outcome. The CRQ Fatigue Domain has a range of 1 to 7, with higher scores associated with better outcome. The CRQ Mastery Domain has a range of 1 to 7, with higher scores associated with better outcome. The CRQ Emotional Function Domain has a range of 1 to 7, with higher scores associated with better outcome.
Time Frame: 6 months
Population: Only patient participants completed this instrument.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants
Number analyzed (Participants) | 14 | 15
Units on a Scale
  CRQ Dyspnea Domain | 4.0 (1.7) | 3.9 (1.7)
  CRQ Fatigue Domain | 3.4 (1.7) | 3.5 (1.5)
  CRQ Mastery Domain | 5.0 (1.4) | 4.5 (1.5)
  CRQ Emotional Function Domain | 4.7 (1.7) | 4.9 (1.6)

7. Secondary Outcome: PROMIS Global Health 10
Description: The PROMIS Global Health 10 is a 10-item measure of quality of life along 2 domains: physical and mental health. There are 9 questions rated on a 5-point Likert-scale, and the 10th question rates pain on a scale of 0 to 10. Raw scores are then converted to standardized t-scores ranging from 0 to 100, with lower scores associated with worse quality of life. PROMIS Global Health Physical Health Domain has a range of 0 to 100, with lower scores associated with worse quality of life. The PROMIS Global Health Mental Health Domain has a range of 0 to 100, with lower scores associated with worse quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 8 | 10
Units on a Scale
  PROMIS Global Health - Physical Health Domain | 36.5 (6.1) | 35.5 (8.3) | 52.2 (8.9) | 51.1 (5.5)
  PROMIS Global Health - Mental Health Domain | 45.8 (8.3) | 40.5 (9.7) | 56.6 (5.7) | 56.0 (8.7)

8. Secondary Outcome: Montgomery Borgatta Caregiver Burden
Description: 14-item measure of caregiver burden along 3 domains: objective burden (alpha=0.87-0.90; Range 6 to 30), subjective stress burden (alpha=0.81-0.88; Range 4 to 20), and subjective demand burden (alpha =0.68-0.82; Range 4 to 20). Higher scores are associated with worse outcome on each domain.
Time Frame: 6 months
Population: Only caregiver participants were included in the analysis of this outcome.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Intervention (EPIC + Usual Care): Caregiver Participants: Caregiver participants randomized to the intervention arm alongside the patient participant receive the caregiver-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, alongside usual care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults and their caregivers. The caregiver-focused EPIC intervention includes four once weekly telephone-based, nurse coach-led sessions tailored to caregivers of patients with COPD aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions and complete an Advance Directive.
Arm/Group | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 8 | 10
Units on a scale
  Objective Burden Domain | 19.3 (2.4) | 20.9 (3.4)
  Subjective Stress Burden Domain | 12.4 (0.9) | 12.9 (1.9)
  Subjective Demand Burden Domain | 11.5 (1.7) | 12.1 (1.8)

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: 14-item measure of emotional symptoms with a 7-item anxiety subscale and a 7-item depression subscale. Each question has a 4-point Likert scale, and scores from 0-21 per subscale, with higher scores associated with more severe anxiety and depressive symptoms. A subscale score >=8 on each subscale is the accepted threshold for clinically-elevated anxiety or depressive symptoms. The minimal clinically important difference is 1.5 points on each subscale with an alpha=0.82-0.83.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Intervention (EPIC): Caregiver Participants: Caregiver participants randomized to the intervention arm alongside the patient participant receive the caregiver-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, alongside usual care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults and their caregivers. The caregiver-focused EPIC intervention includes four once weekly telephone-based, nurse coach-led sessions tailored to caregivers of patients with COPD aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions and complete an Advance Directive.
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 8 | 10
Units on a scale
  HADS Depression Subscale | 6.4 (3.3) | 8.3 (5.3) | 2.5 (1.9) | 2.6 (1.7)
  HADS Anxiety Subscale | 5.1 (3.2) | 6.6 (4.3) | 2.5 (1.8) | 3.4 (2.2)

10. Secondary Outcome: Modified Telephone Interview for Cognitive Status (mTICS)
Description: 14-item measure of cognitive impairment, which has been validated in COPD. Scores range from 0-50 with higher scores associated with more cognitive impairment. Validated over telephone (alpha=0.80).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Intervention (): Patient Participants: Patient participants randomized to the intervention arm receive the patient-focused EPIC (Empower People to Independence in COPD) intervention, a telephonic nurse coach-led palliative care intervention informed by the ENABLE (Educate, Nurture, Advise, Before Life Ends) model for early palliative care, alongside usual care. ENABLE is a rigorously tested multicomponent early palliative care model that improved quality of life and emotional symptoms in patients with advanced cancer. The PI adapted and refined ENABLE for COPD and older adults. The patient-focused EPIC intervention includes six once weekly telephone-based, nurse coach-led sessions aided by a manualized curriculum (Charting Your Course), followed by three once-monthly follow up sessions. Participants also complete activities on solving problems and making difficult decisions, complete an Advance Directive, and attend a supportive care clinic visit. Caregiver participants are randomized to the same study arm as the patient participant and receive the caregiver-focused EPIC intervention with four caregiver-tailored nurse-coach sessions, instead of six sessions.
Arm/Group | Intervention (): Patient Participants | Control (Usual Care): Patient Participants
Number analyzed (Participants) | 13 | 15
Units on a scale | 28.6 (4.4) | 31.7 (6.6)

11. Secondary Outcome: Katz Index of Activities of Daily Living
Description: 6-item measure of independence in activities. Range 0-6. Higher scores associated with more independence; MCID=0.47.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention (): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 8 | 10
Units on a scale | 5.7 (0.7) | 5.3 (1.6) | 6.0 (0.0) | 6.0 (0.0)

12. Secondary Outcome: Lawton Instrumental Activities of Daily Living
Description: 8-item measure of function in independent living, with an MCID=0.47. Scores range from 1 to 8, with higher scores associated with higher functioning. alpha=0.85
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 8 | 10
Units on a scale | 5.0 (2.0) | 5.7 (1.8) | 7.0 (1.4) | 7.7 (1.9)

13. Secondary Outcome: Advance Directive Completion
Description: Rates of patient participant Advance Directive completion.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants
Number analyzed (Participants) | 14 | 15
Participants | 7 | 5

14. Secondary Outcome: De Jon Gierveld Loneliness Scale
Description: A 6-item measure of loneliness with higher scores associated with more loneliness, range 0 (least lonely) to 6 (most lonely). Alpha=0.88.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Control (Usual Care): Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Control (Usual Care): Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 8 | 10
Units on a scale | 1.8 (1.4) | 2.6 (2.1) | 1.1 (1.6) | 0.8 (1.3)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Usual Care: Patient Participants: Participants randomized to this arm will receive the standard of care for COPD.
  Usual COPD Care: Participants randomized to this arm receive standard of care for COPD. This includes routine clinic visits with their clinician, medications, inhalers, vaccinations, tobacco cessation counseling, illness education, cardiopulmonary rehabilitation, specialist referrals, and other COPD therapies deemed appropriate by their clinician.
- Usual Care: Caregiver Participants: Participants randomized to this arm will receive usual care.
Arm/Group | Intervention (EPIC + Usual Care): Patient Participants | Usual Care: Patient Participants | Intervention (EPIC + Usual Care): Caregiver Participants | Usual Care: Caregiver Participants
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT05040386/Prot_SAP_000.pdf